CLINICAL TRIAL: NCT01215136
Title: Phase II Trial of Everolimus or Everolimus Plus Paclitaxel as First-line Therapy in Cisplatin-ineligible Patients With Advanced Urothelial Carcinoma: Hoosier Cancer Research Network GU10-147
Brief Title: First-line Everolimus +/- Paclitaxel for Cisplatin-ineligible Patients With Advanced Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Matthew Galsky (Other)
Collaborators: Hoosier Cancer Research Network (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU10-147
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Transitional Cell Carcinoma; Bladder Carcinoma; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Everolimus; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Active Comparator): Single-agent everolimus (enrollment limited to patients with patients with creatinine clearance < 60 ml/min AND Karnofsky performance status of 60-70%)
  Interventions: Drug: Everolimus
- Cohort 2 (Active Comparator): Everolimus plus paclitaxel (enrollment limited to patients with creatinine clearance < 60 ml/min OR Karnofsky performance status of 60-70%)
  Interventions: Drug: Everolimus; Drug: Paclitaxel

INTERVENTIONS:
Drug: Everolimus — 10 mg PO daily (continuously, without scheduled treatment interruptions). The cycle length will last 28 days. Everolimus will be dispensed on Day 1 of each cycle by the study center personnel on an outpatient basis.
  Arms: Cohort 1
Drug: Everolimus — 10 mg PO daily (continuously, without scheduled treatment interruptions). The cycle length will last 28 days. Everolimus will be dispensed on Day 1 of each cycle by the study center personnel on an outpatient basis.
  Arms: Cohort 2
Drug: Paclitaxel — Paclitaxel 80 mg/m2 IV as a 1 hour infusion on days 1, 8, and 15, of a 28-day cycle.
  Arms: Cohort 2

SUMMARY:
The purpose of this trial is to explore the activity and safety of everolimus +/- paclitaxel as first-line therapy for cisplatin-ineligible patients with advanced urothelial carcinoma.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study

Patients will be enrolled into one of two parallel cohorts:

* Cohort 1: impaired renal function AND poor performance status (cycle length = 28 days). Everolimus 10 mg orally daily
* Cohort 2: impaired renal function OR poor performance status (cycle length = 28 days). Everolimus 10 mg orally daily + IV Paclitaxel 80 mg/m2 on D1, 8, 15

Restaging evaluations will be performed after every 2 cycles.

Treatment will continue until disease progression or unacceptable toxicity.

Karnofsky performance status 60-70%

Life Expectancy: Not specified

Hematopoietic:

* Absolute neutrophil count (ANC) ≥ 1.5 K/mm3
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets ≥ 100 K/mm3
* INR ≤ 1.5 (Anticoagulants are allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of Low molecular weight (LMW) heparin for at least 2 weeks prior to registration for protocol therapy).
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L
* Fasting triglycerides ≤ 2.5 x ULN.
* Fasting serum glucose < 1.5 x ULN

Hepatic:

* Bilirubin ≤ 1.5 x ULN
* Aminotransferases (AST and ALT) ≤ 2.5 x ULN (unless liver metastases, then ≤ 5 x ULN)

Renal:

* Calculated creatinine clearance of < 60 using the Cockcroft-Gault formula

Cardiovascular:

* No symptomatic congestive heart failure of New York heart Association Class III or IV.
* No unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of transitional cell carcinoma (TCC) of the bladder, urethra, ureter, or renal pelvis (urothelial carcinoma). Histology may be mixed, but still requires a component of TCC.
* Measurable disease according to RECIST and obtained by imaging within 30 days prior to registration for protocol therapy.
* Must be ineligible for cisplatin, based on the following, within 30 days prior to registration for protocol therapy.
* Prior radiation therapy is allowed to < 25% of the bone marrow.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years at the time of consent.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 8 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to prior to registration for protocol therapy.
* Females must not be breastfeeding.

Exclusion Criteria:

* No prior chemotherapy for metastatic disease. Prior chemotherapy in the neoadjuvant/adjuvant setting is allowed if completed at least 12 months prior to registration for protocol therapy.
* No active CNS metastases or leptomeningeal metastases. Patients with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis.
* No prior malignancy is allowed except for adequately treated basal cell or adequately treated squamous cell skin cancer, in situ cervical cancer, Gleason ≤ grade 7 prostate cancers (treated definitively with no evidence of PSA progression), or other cancer for which the patient has been disease-free for at least 5 years.
* No treatment with any anticancer therapy or investigational agent within 30 days prior to registration for protocol therapy.
* No known hypersensitivity to any protocol treatment.
* No prior treatment with mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* No history of immunization with attenuated live vaccines within one week prior to registration for protocol therapy or during study period.
* No severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air.
* No uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN.
* No active (acute or chronic) or uncontrolled severe infections.
* No liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
* No known history of HIV seropositivity.
* No impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* No active, bleeding diathesis.
* No history of major surgery (defined as requiring general anesthesia) or significant traumatic injury within 30 days prior to registration for protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-12; Primary Completion 2017-04-24 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, M.D., Study Chair — Hoosier Cancer Research Network
Locations (11):
- United States (11):
  - University of Alabama Hematology Oncology Clinic at Medical West, Birmingham, Alabama
  - Northwestern University, Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - Metro Health Cancer Care, Wyoming, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Icahn School of Medicine: Tisch Cancer Institute at Mount Sinai Medical Center, New York, New York
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

REFERENCES:
- [Derived] Jun T, Hahn NM, Sonpavde G, Albany C, MacVicar GR, Hauke R, Fleming M, Gourdin T, Jana B, Oh WK, Taik P, Wang H, Varadarajan AR, Uzilov A, Galsky MD. Phase II Clinical and Translational Study of Everolimus +/- Paclitaxel as First-Line Therapy in Cisplatin-Ineligible Advanced Urothelial Carcinoma. Oncologist. 2022 Jun 8;27(6):432-e452. doi: 10.1093/oncolo/oyab075. PMID 35438782
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus: Single-agent everolimus (enrollment limited to patients with patients with creatinine clearance < 60 ml/min AND Karnofsky performance status of 60-70%)
  Everolimus: 10 mg PO daily (continuously, without scheduled treatment interruptions). The cycle length will last 28 days. Everolimus will be dispensed on Day 1 of each cycle by the study center personnel on an outpatient basis.
- Everolimus Plus Paclitaxel: Everolimus plus paclitaxel (enrollment limited to patients with creatinine clearance < 60 ml/min OR Karnofsky performance status of 60-70%)
  Everolimus: 10 mg PO daily (continuously, without scheduled treatment interruptions). The cycle length will last 28 days. Everolimus will be dispensed on Day 1 of each cycle by the study center personnel on an outpatient basis.
  Paclitaxel: Paclitaxel 80 mg/m2 IV as a 1 hour infusion on days 1, 8, and 15, of a 28-day cycle.
Period: Overall Study
Arm/Group | Everolimus | Everolimus Plus Paclitaxel
Started | 7 | 29
Completed | 1 | 2
Not Completed | 6 | 27
Not completed — Adverse Event | 2 | 9
Not completed — Disease Progression | 3 | 14
Not completed — Symptomatic Deterioration | 1 | 1
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Everolimus Plus Paclitaxel | Total
Number analyzed (Participants) | 7 | 29 | 36
Age, Continuous [Mean (Full Range); unit: years] | 78 [59 to 90] | 72.14 [54 to 88] | 73.28 [54 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 5 | 22 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 28 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 5 | 27 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 29 | 36
Karnovsky Performance Status (KPS) at Screening [Count of Participants; unit: Participants] — KPS is a general indicator of a subject's well being and ability to carry on daily activities.
  100:Normal no complaints 90:Able to carry on normal activity 80:Normal activity with effort; some signs or symptoms of disease. 70:Cares for self 60:Requires occasional assistance, but is able to care for most of his personal needs. 50:Requires considerable assistance and frequent medical care.
  40:Disabled 30:Severely disabled 20:Very sick 10:Moribund 0:Dead
  Participants
    KPS 100 | 0 | 4 | 4
    KPS 90 | 0 | 6 | 6
    KPS 80 | 0 | 12 | 12
    KPS 70 | 1 | 4 | 5
    KPS 60 | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Single-Agent Everolimus and Everolimus + Paclitaxel
Description: To evaluate clinical benefit rate (complete response, partial response, and stable disease) at 4 months from initiation of treatment.
Time Frame: 4 months
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 29
percentage of participants | 14.3 | 37.9

2. Secondary Outcome: Number of Adverse Events as a Measure of Safety and Tolerability
Description: To determine the safety of everolimus and everolimus plus paclitaxel in this patient population. A summary with the count of events per grade is provided.
Time Frame: 5 months
Measure: Number; unit: Number of Events
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 29
Number of Events
  Grade 1 Adverse Events | 10 | 116
  Grade 2 Adverse Events | 9 | 75
  Grade 3 Adverse Events | 4 | 39
  Grade 4 Adverse Events | 0 | 1
  Grade 5 Adverse Events | 0 | 3

3. Secondary Outcome: Progression Free Survival
Description: To determine median progression free survival per RECIST 1.1, per cohort.
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 29
months | 2.3327 [1.6099 to 3.5483] | 5.8480 [2.9569 to 7.6550]

4. Secondary Outcome: Overall Survival
Description: To determine median overall survival at 1-year from the initiation of treatment.
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 29
months | 4.5010 [2.2341 to 8.3121] | 10.8747 [6.8337 to 14.3573]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 12 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored for up to 5 months.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 7/7 | 25/29
Serious Adverse Events (participants affected / at risk) | 1/7 | 11/29
Other Adverse Events (participants affected / at risk) | 5/7 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=29)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (1) | 2 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
EDEMA LIMBS (General disorders) | 0 (0) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=29)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 2 (5) | 17 (73)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (3) | 11 (23)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 6 (6)
FATIGUE (General disorders) | 3 (3) | 15 (29)
FEVER (General disorders) | 1 (1) | 4 (5)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (6) | 14 (25)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 10 (11)
PERINEAL PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (14)
VOMITING (Gastrointestinal disorders) | 1 (1) | 4 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 13 (19)
AORTIC VALVE DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 1 (1)
CHOLESTEROL HIGH (Investigations) | 0 (0) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 3 (4)
CREATININE INCREASED (Investigations) | 0 (0) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2)
DRY EYE (Eye disorders) | 0 (0) | 1 (1)
EDEMA LIMBS (General disorders) | 0 (0) | 6 (9)
EDEMA TRUNK (General disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
HAPTOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1)
HEAD SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 0 (0) | 7 (9)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 0 (0) | 2 (2)
INSOMNIA (Psychiatric disorders) | 0 (0) | 3 (3)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NAIL INFECTION (Infections and infestations) | 0 (0) | 2 (4)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 9 (19)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
PELVIC INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 11 (13)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 6 (16)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1)
SALIVARY GLAND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 1 (1)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 5 (5)
WEIGHT LOSS (Investigations) | 0 (0) | 4 (7)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT01215136/Prot_SAP_000.pdf